CLINICAL TRIAL: NCT00487279
Title: DEfibrillators To REduce Risk by MagnetIc ResoNance Imaging Evaluation
Acronym: DETERMINE
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Study terminated early due to inability to enroll.
Sponsor: Abbott Medical Devices (Industry)
Collaborators: Northwestern University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Determine2007v12
Record Dates: First submitted 2007-06-13; First posted 2007-06-18 (Estimated); Results first posted 2012-03-26 (Estimated); Last update posted 2019-02-05 (Actual); Status verified 2019-02

CONDITIONS: Coronary Artery Disease; Left Ventricular Dysfunction; Sudden Cardiac Death
Keywords: Coronary; Artery; Disease; Sudden; Cardiac; Death; ICD
MeSH Terms: conditions — Coronary Artery Disease; Ventricular Dysfunction, Left; Death, Sudden, Cardiac; Disease; Death | interventions — Defibrillators; Defibrillators, Implantable

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- ICD Group (Experimental): ICD (Implantable Cardioverter Defibrillator)
  Interventions: Device: Defibrillator
- Control Group (Other): Medial Therapy
  Interventions: Other: Control

INTERVENTIONS:
Device: Defibrillator — ICD(Implantable Cardioverter Defibrillator)
  Other Names: Implantable Cardioverter Defibrillator
  Arms: ICD Group
Other: Control — No Intervention
  Other Names: No Intervention
  Arms: Control Group

SUMMARY:
This trial is a prospective, multi-center, randomized study of patients with coronary artery disease (CAD) and mild to moderate left ventricular (LV) dysfunction. The primary objective of this study is to test the hypothesis that Implantable Cardioverter Defibrillator (ICD) therapy in combination with medical therapy in patients with an infarct size greater than or equal to 10% of the left ventricular mass improves long term survival compared to medical therapy alone. In addition to the 2-arm randomized trial, the study will also include a non-investigational registry of non-randomized patients.

DETAILED DESCRIPTION:
Detailed Description:

The utilization of ICD therapy has resulted in significant reduction in mortality among those at highest risk of sudden cardiac death, such as survivors of cardiac arrest and patients presenting with symptomatic sustained ventricular arrhythmias. Patients with CAD and advanced LV dysfunction (EF <35%) also benefit from ICD. However, although at high risk, these patients represent only a small percentage of the population who die suddenly. While there are many tests that have been used for stratification of risk for sudden cardiac death, the two that have documented clinical utility are determination of left ventricular ejection fraction and presence of inducibility of ventricular tachycardia during programmed electrical stimulation performed as part of EP testing. The utility of these tests likely result from their ability to select patients who have the requisite substrate allowing for sustained ventricular tachyarrhythmias. It has been shown that ventricular tachycardia occurs more commonly in the setting of larger infarcts. Ejection fraction has been related to infarct size; presumably, the larger the area of infarction, the lower the ejection fraction. Electrophysiologic testing directly establishes the presence of substrate by the actual induction of ventricular tachycardia.

A major limitation of electrophysiologic programmed stimulation is the high number of false negative findings. Thus, a significant number of patients without inducible arrhythmias remain at risk. CE-MRI provides functional information (EF, LV Volumes, LV mass, etc), which is routine in the initial evaluation of post-MI patients, and in addition provides detailed geometry of scar tissue. There is a clear association between inducible arrhythmias and scar size which until the development of cardiac MRI, could not be seen in humans. Use of cardiac MRI has demonstrated that although most patients with a large MI were inducible, a small but significant number of patients, who remain at risk, were not inducible. There was also an association between death and infarct size in patients with cardiovascular risk factors but no established CAD.

The Center for Medicare Services (CMS) has recently decided in a coverage decision that patients with left ventricular dysfunction, heart failure, and an ejection fraction of <35% would be eligible to receive an ICD as long as they are enrolled in a prospective registry. Patients with LV ejection fractions greater than 35% or those without heart failure and ejection fractions over 30%, represent a more difficult management dilemma. However, since the majority of out of hospital cardiac arrests occur in patients with EF >35%, managing these patients is crucial in addressing the epidemiologic problem of sudden cardiac death.

The primary objective of this trial is to test the hypothesis that therapy with an ICD combined with medical therapy improves long-term survival compared to medical therapy alone in patients with CAD, infarct mass greater than or equal to 10% of the left ventricle and left ventricular dysfunction who do not have an indication for ICD by either of the following criteria. Patients must have an EF of >35% or have an EF of 30-35% and must not have inducible ventricular tachycardia or have NYHA Class II or greater heart failure (Target Population).

The secondary objective is to test the hypothesis that therapy with an ICD combined with medical therapy improves arrhythmic survival compared to medical therapy alone in patients with CAD, infarct mass greater than or equal to 10% and left ventricular dysfunction who do not have an indication for ICD based on the Target Population described above.

Recruitment: All patients who have a history of coronary heart disease (CAD) with documentation of either myocardial infarction (MI) or left ventricular dysfunction (LVD), a preliminary ejection fraction (EF) > 35% and have previously undergone a contrast-enhanced MRI (CE-MRI) study for clinical diagnostic reasons or as part of the study entry screening procedure may be further evaluated for eligibility for this trial. In addition, patients with an ejection fraction of 30-35% may be eligible for the study if they do not currently have an indication for an ICD based on Target Population criteria described above. These patients may have NYHA Class I heart failure, no non-sustained VT on holter monitor, or if non-sustained VT is present, there is the absence of inducible VT at EP study.

The first 1550 patients who are found to have an EF >30% with NYHA Class I heart failure or 35% by routine clinical evaluation and who also have an MI involving greater than or equal to 10% of total left ventricular mass will be enrolled in the main randomized portion of the trial. These patients will be randomly assigned to one of two groups: ICD therapy in combination with medical therapy (ICD Group) or medical therapy alone (Control Group).

Follow-Up: Clinic visits are required every 6 months until the completion of the study. Telephone contact is required every six months to assess vital status and obtain new information regarding medical status and/or medical events. The telephone calls alternate with the clinical visits, so that patient contact will occur every 3 months until the completion of the study.

Non-Investigational Registry:

The primary objective of the registry sub-study is to test the hypothesis that infarct mass as measured by contrast enhanced Cardiac MRI (CE-MRI) is a better predictor for sudden cardiac death than LV ejection fraction. The registry will examine infarct mass as measured by Cardiac MRI and LV ejection fraction (EF) as predictors for SCD.

The purpose of the registry is hypothesis generating and no labeling or other indications are anticipated based on registry findings.

Participation in the Registry requires that the patient has undergone a contrast-enhanced cardiac MRI prior to enrollment. In order to ensure consistent infarct mass assessments, the cardiac MRI study submitted to determine eligibility for randomization must meet the following criteria:

1. CE-cardiac MRIs must be obtained using Siemens, General Electric or Phillips equipment.
2. The contrast agent must be gadolinium-based at a dose sufficient to render images of acceptable quality.
3. The CE-cardiac MRI must be available for electronic submission to the MRI Core laboratory for analysis.

If techniques for infarct mass measurement or data acquisition change during the course of the trial, the Core laboratory and the Steering Committee may choose to alter some of the above parameters.

Once consent to participate in the registry has been obtained, the site will forward the CE-MRI study to the CE-MRI core lab for analysis to determine placement in the appropriate registry, baseline demographics characteristics will be collected on all registry patients. This will aid in statistical analysis to verify the generalizability of the findings. The differences in total survival between these groups will also be compared using the same methodology as for the primary end-point. Patients with and without ICD implants will be compared separately. In addition, blood specimens for genetic sampling and biomarker testing will be obtained on all patients in the registry cohort who agree, to determine if any of SCD substrates exist in the DETERMINE registry population.

Study subjects will be contacted by mail by the Endpoint Coordinating Center at Brigham and Women's Hospital in Boston every 6 months to determine vital status and obtain any new information regarding change in medical status or the occurrence of any medical events. This will promote the continued relationship between the study participant and the enrolling center and can also be used to remind the study subject of their next scheduled appointment.

Scope and Duration of the trial:

* Up to 100 sites to screen a total of 10,000 patients will enroll 1550 patients into the randomized study recruited from a total of 10,000 patients contributing data and CE-MRI images to the registries.
* Registry enrollment per site = ~90 subjects
* Randomization per site = 1-3 per month (expected randomized enrollment per site is 20 patients or more )
* Estimated enrollment period: 36 months
* 24 months of follow-up after the last patient is randomized

ELIGIBILITY:
Inclusion Criteria:

Randomized Arm

1. Evidence of Coronary Artery Disease (CAD)a.
2. Evidence of prior Myocardial Infarction defined by either:

   A. Clinical history of prior myocardial infarction OR B. Mild-moderate systolic LV dysfunction with an EF ≤50%
3. LVEF>35% by any current standard evaluation technique (e.g., echocardiogram, MUGA, angiography).

   • Patients who have an EF between 30-35% and NYHA Class I heart failure who do not have a history of ventricular tachyarrhythmias, or inducible ventricular tachycardia during electrophysiological (EP) testing can be enrolled (Target Population).
4. CE-MRI measure of infarct mass > 10% of LV mass (as measured by the MRI core lab)

   • If CE-MRI performed ≤ 40 days after myocardial infarction infarct mass must be ≥ 15% of the LV mass.
5. Patients aged 18 years or above

   1. CAD will be confirmed by evidence of one of the following three (3) criteria 1) Prior myocardial infarction, 2) Significant stenosis of a major epicardial vessel (>50% proximal or 70% distal) by coronary angiography, 3) Prior revascularization (percutaneous coronary intervention or coronary artery bypass surgery. Patients may not be randomized until 90 days after revascularization.
   2. MI should be documented by the presence of two (2) of the following three (3) criteria: 1) Symptoms consistent with myocardial infarction (i.e. chest pain, shortness of breath), 2) Q-waves on electrocardiogram and 3) Elevated cardiac enzymes (CPK elevation > two times or troponin elevation > three times the upper limit of normal for the lab). Patients may not be randomized until 40 days after myocardial infarction.

Exclusion Criteria

1. History of cardiac arrest or spontaneous or inducible sustained VT (15 beats or more at a rate of 120 BPM or greater)*
2. Unexplained syncope
3. Need for revascularization based on investigator's clinical assessment within the next 12 months (patients may be reevaluated 90 days after revascularization)
4. Currently implanted permanent pacemaker and/or pacemaker/ICD lead
5. Contraindication to a ICD implant (i.e. inadequate venous access, bleeding disorder)
6. Acute or chronic severe renal insufficiency (< 30mL/min/1.73m2); acute renal insufficiency of any severity due to hepato-renal syndrome
7. Current or planned renal or liver transplant
8. End stage renal disease on hemodialysis or peritoneal dialysis
9. Contraindication to CE-MRI or history of allergy to gadolinium-based contrast dye
10. Metal fragments in the eyes or face, implantation of any electronic devices such as (but not limited to) cardiac pacemakers, cardiac defibrillators, cochlear implants or nerve stimulators, surgery on the blood vessels of the brain, body piercing
11. Recent MI (<40 days) or revascularization (<90 days)
12. CVA within 90 days
13. Antiarrhythmic drug therapy for ventricular arrhythmias
14. New York Heart Association CHF functional class IV at enrollment

Non-Investigational Registry Inclusion Criteria

* Evidence of CAD a with either a history of prior myocardial infarction OR any LV dysfunction
* Evidence of LV dysfunction (ejection fraction) as measured by any current standard screening technique (e.g., echocardiogram, MUGA, angiography).c
* Clinical CE-MRI within the past 12 months (scheduled or completed)
* Patients aged 18 years or above
* CAD will be confirmed by evidence of one of the following three (3) criteria 1) Prior myocardial infarction, 2) Significant stenosis of a major epicardial vessel (>50% proximal or 70% distal) by coronary angiography, 3) Prior revascularization (percutaneous coronary intervention or coronary artery bypass surgery.
* MI should be documented by the presence of two (2) of the following three (3) criteria: 1) Symptoms consistent with myocardial infarction (i.e. chest pain, shortness of breath), 2) Q-waves on electrocardiogram and 3) Elevated cardiac enzymes (CPK elevation > two times or troponin elevation > three times the upper limit of normal for the lab).
* Patients can be enrolled in the registry even if they have received or are about to receive an ICD for primary prevention.

Exclusion Criteria

* History of cardiac arrest or spontaneous or inducible sustained VT (15 beats or more at a rate of 120BPM or greater)*
* Contraindication to CE-MRI or history of allergy to gadolinium-based contrast
* Spontaneous arrhythmia that precludes assessment by cardiac MRI
* Acute or chronic severe renal insufficiency (<30mL/min/1.73m2); acute renal insufficiency of any severity due to hepato-renal syndrome.
* Current or planned renal or liver transplant
* End stage renal disease on hemodialysis or peritoneal dialysis
* Metal fragments in the eyes or face, implantation of any electronic devices such as (but not limited to) cardiac pacemakers, cardiac defibrillators, cochlear implants or nerve stimulators, surgery on the blood vessels of the brain , body piercing
* Uninterpretable MRI images by core lab criteria
* Any condition other than cardiac disease that, in the investigator's judgment, would seriously limit life expectancy (poor 6-month survival)
* Marked valvular heart disease requiring surgical intervention
* Current alcohol or drug abuse
* Participating in other trials with an active treatment arm (not to exclude patients who are in trials of diagnostic techniques or approved therapies)
* Unwilling or unable to provide informed consent *Exception: Cardiac arrest or spontaneous VT that occurs during the acute MI event will not be considered an exclusion

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 81 (Actual)
Dates: Start 2007-06; Primary Completion 2010-12 (Actual); Study Completion 2011-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Alan Kadish, MD, Principal Investigator — Northwestern University
Locations (56):
- United States (56):
  - Alaska Regional Hospital and Alaska Cardiovascular Research Foundation, LLC, Anchorage, Alaska
  - University of Arizona, Tucson, Arizona
  - Glendale Memorial Hospital and Health Center, Glendale, California
  - Long Beach Memorial Medical Center, Long Beach, California
  - Hollywood Presbyterian Medical Center, Los Angeles, California
  - UCLA Medical Center, Los Angeles, California
  - Hoag Memorial Hospital Presbyterian and Radin Inc., Newport Beach, California
  - Catholic Healthcare West (d/b/a mercy General Hospital) and Regional Cardiology Associates, Sacramento, California
  - Rocky Mountain Cardiovascular Associates, Denver, Colorado
  - University of Florida-Shands/Jacksonville, Jacksonville, Florida
  - Orlando Regional Healthcare System, Orlando, Florida
  - Cardiology Consultants of Northwest Florida, Pensacola, Florida
  - Emory University, Atlanta, Georgia
  - Northeast Georgia Heart Center, PC, Gainesville, Georgia
  - Northwestern University, Chicago, Illinois
  - Midwest Heart Foundation, Lombard, Illinois
  - Lutheran Hospital of Indiana and Northern Indiana Research Alliance of the Heart Center Medical Group, Fort Wayne, Indiana
  - The Care Group, Indianapolis, Indiana
  - Kentucky Heart Institute / King's Daughter, Ashland, Kentucky
  - Baptist Healthcare System Inc. (d/b/a Central Baptist Hospital), Lexington, Kentucky
  - Johns Hopkins, Baltimore, Maryland
  - MedStar Research Institute (Washington Hospital Center), Hyattsville, Maryland
  - The Brigham and Women's Hospital Inc., Boston, Massachusetts
  - Caritas St. Elizabeth's Medical Center, Boston, Massachusetts
  - Henry Ford Health System, Detroit, Michigan
  - Advanced Cardiac Healthcare (Bronson Methodist Hospital), Kalamazoo, Michigan
  - William Beaumont Hospital, Royal Oak, Michigan
  - Minneapolis Heart Institute Foundation/Abbott NW Hospital, Minneapolis, Minnesota
  - Metropolitan Cardiology Consultants (MCC) / Allina Health System (Mercy & Unity Hospitals), Minneapolis, Minnesota
  - University of Nebraska Medical Center, Omaha, Nebraska
  - Valley Hospital, Ridgewood, New Jersey
  - New York Methodist Hospital, Brooklyn, New York
  - St. Luke's - Roosevelt Hospital Center, New York, New York
  - Columbia University Medical Center, New York, New York
  - University of Rochester, Rochester, New York
  - St. Francis Hospital, Roslyn, New York
  - LeBauer Cardiovascular Research Foundation and Moses H. Cone Memorial Hospital, Greensboro, North Carolina
  - University of Maryland Baltimore and Maryland Medical Center, Cleveland, Ohio
  - University Hospitals of Cleveland, Cleveland, Ohio
  - MetroHealth Medical Center, Cleveland, Ohio
  - The Cleveland Clinic Foundation, Cleveland, Ohio
  - North Ohio Research, Ltd., Elyria, Ohio
  - AHS Hillcrest Medical Center, LLC and Oklahoma Heart Institute, Tulsa, Oklahoma
  - Abington Memorial Hospital, Abington, Pennsylvania
  - Lehigh Valley Hospital and Health Network, Allentown, Pennsylvania
  - Allegheny-Singer Research Institute, Pittsburgh, Pennsylvania
  - University of Pittsburgh Medical Center, Pittsburgh, Pennsylvania
  - Stern Cardiovascular Center, Germantown, Tennessee
  - Centennial Medical Center, Nashville, Tennessee
  - St. Thomas Research Institute, LLC, Nashville, Tennessee
  - Vanderbilt Medical Center, Nashville, Tennessee
  - Methodist Hospital Research Institute, Houston, Texas
  - St. Luke's Episcopal Hospital, Houston, Texas
  - Sentara Hospitals and Sentara Cardiovascular Research Institute, Norfolk, Virginia
  - Cardiovascular Associates Virginia Beach, Virginia Beach, Virginia
  - North Cascade Cardiology, Bellingham, Washington

RESULTS

PARTICIPANT FLOW:
Groups:
- ICD Group: ICD (Implantable Cardioverter Defibrillator)in combination with medical therapy
- Control Group: Medical therapy alone
Period: Overall Study
Arm/Group | ICD Group | Control Group
Started | 44 | 37
Completed | 43 | 35
Not Completed | 1 | 2
Not completed — Death | 1 | 0
Not completed — Withdrawal by Subject | 0 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | ICD Group | Control Group | Total
Number analyzed (Participants) | 44 | 37 | 81
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 24 | 16 | 40
  >=65 years | 20 | 21 | 41
Age, Continuous [Mean (Standard Deviation); unit: years] | 62 (11) | 65 (12) | 63 (12)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11 | 5 | 16
  Male | 33 | 32 | 65
Region of Enrollment [Number; unit: participants]
  United States | 44 | 37 | 81

OUTCOME MEASURES:

1. Primary Outcome: All-cause Mortality
Time Frame: Total survival will be evaluated 2 years after the last patient is randomized.
Population: Intent to Treat
Measure: Number; unit: participants
Arm/Group | ICD Group | Control Group
Number analyzed (Participants) | 44 | 37
participants | 1 | 0

2. Secondary Outcome: Arrhythmic Mortality
Description: Arrhythmic mortality was reported as the number of randomized patients who died due to arrhythmic death. Arrhythmic death was defined as death due to arrhythmia or sudden death.
Time Frame: Total survival will be evaluated 2 years after the last patient is randomized.
Measure: Number; unit: participants
Arm/Group | ICD Group | Control Group
Number analyzed (Participants) | 44 | 37
participants | 0 | 0

ADVERSE EVENTS:
Description: Serious adverse events were defined as those related to the device or its implantation procedure. Therefore, the control group was not at risk for a serious adverse event. Other adverse events were defined as non-serious adverse events related to the ICD or its implant procedure. The control group was not at risk for an other adverse event.
Arm/Group | ICD Group | Control Group
Serious Adverse Events (participants affected / at risk) | 3/44 | 0/0
Other Adverse Events (participants affected / at risk) | 2/44 | 0/0
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs (number of events):
Term (organ system) | ICD Group (N=44) | Control Group (N=0)
Lead Dislodgment or Migration (Injury, poisoning and procedural complications) | 3/3 (3) | 0 (0) — Serious adverse events were defined as those events related to the device or its implantation. Therefore the control group was not at risk for a serious adverse event per the protocol definition.
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs (number of events):
Term (organ system) | ICD Group (N=44) | Control Group (N=0)
Infection (Infections and infestations) | 1/1 (1) | 0 (0)
Lead Dislodgment or Migration (Injury, poisoning and procedural complications) | 1/1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
All publications must be reviewed by the Sponsor, Executive Sterring Committe and the Publications Committee at least 30 days prior to submittal. In the event that no multi-center study publication occurs within 12 months of study completion, investigators may publish the restuls of the study data from those subjects enrolled in a study at the Institution provided the Sponsor, Executive Steering Committee and Publicaiton Committee review at least 30 days prior to submittal.